CLINICAL TRIAL: NCT00058396
Title: Phase I Study Of IDEC-152 (Anti-CD23 Monoclonal Antibody) In Patients With Relapsed Or Refractory Chronic Lymphocytic Leukemia
Brief Title: Monoclonal Antibody in Treating Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: IDEC-152-20; MSKCC-02096; CDR0000288828 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2009-12

CONDITIONS: Leukemia; Lymphoma
Keywords: refractory chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; noncontiguous stage II small lymphocytic lymphoma; recurrent small lymphocytic lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; contiguous stage II small lymphocytic lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — lumiliximab

INTERVENTIONS:
Biological: lumiliximab

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of monoclonal antibody therapy in treating patients who have relapsed or refractory chronic lymphocytic leukemia or small lymphocytic lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine a recommended phase II dose of IDEC-152 monoclonal antibody in patients with relapsed or recurrent chronic lymphocytic leukemia.
* Determine the safety profile of this drug in these patients.
* Determine the pharmacokinetics and pharmacodynamics of this drug in these patients.
* Determine the efficacy of this drug in these patients.

OUTLINE: This is an open-label, multicenter, dose-escalation study.

Patients receive IDEC-152 monoclonal antibody IV over at least 2 hours on days 1, 2, 8, 15, and 22.

Cohorts of 3-10 patients receive escalating doses of IDEC-152 monoclonal antibody until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3, 2 of 6, or 3 of 10 patients experience dose-limiting toxicity.

Patients are followed every 3 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 15-50 patients will be accrued for this study within 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed chronic lymphocytic leukemia OR small lymphocytic lymphoma

  * Stage III-IV OR
  * Stage I-II, if determined to have disease progression evidenced by 1 of the following characteristics:

    * Rapid doubling of peripheral lymphocyte count
    * Progressive lymphadenopathy
    * Progressive splenomegaly
    * B symptoms
    * Grade 2 or 3 fatigue
* CD23+ disease
* Progressive disease after at least 1 prior chemotherapy course

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* At least 6 months

Hematopoietic

* Platelet count at least 50,000/mm^3

Hepatic

* Bilirubin no greater than 2.0 mg/dL
* AST/ALT no greater than 1.5 times upper limit of normal (ULN)

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* No New York Heart Association class III or IV cardiac disease
* No myocardial infarction within the past 6 months
* No unstable arrhythmia
* No evidence of ischemia on EKG within the past 14 days

Pulmonary

* FEV_1 at least 60% of predicted
* DLCO at least 55% of predicted

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study treatment
* HIV negative
* No secondary malignancy requiring active treatment (except hormonal therapy)
* No serious nonmalignant disease that would preclude study participation
* No active uncontrolled bacterial, viral, or fungal infection
* No clinically active autoimmune disease

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior anticancer biologic therapy
* More than 4 weeks since prior anticancer radioimmunotherapy
* No prior exposure to IDEC-152 or anti-CD23 antibodies

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior anticancer chemotherapy

Endocrine therapy

* Concurrent hormonal therapy allowed for second malignancy

Radiotherapy

* More than 4 weeks since prior anticancer radiotherapy

Surgery

* More than 4 weeks since prior major surgery (except for diagnostic surgery)

Other

* More than 4 weeks since prior anticancer investigational therapy
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10; Primary Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Adam Weiss, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States